CLINICAL TRIAL: NCT01489384
Title: A Canadian Randomized Controlled Trial of DMARD Withdrawal in RA Patients Achieving Therapeutic Response With Cimzia + DMARD Combination Treatment.
Brief Title: Cimzia Treatment in Rheumatoid Arthritis: Randomizing to Stop Versus Continue Disease-modifying Anti-rheumatic Drug(s)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pope Research Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PRC-06-2011; JSS-01-2013 (Other: UCB Canada)
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; DAS28
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 3 months: Discontinue vs continue DMARDS: At 3 months those patients who achieved a change in DAS28 of 1.2 or greater will be randomized to discontinue versus continue DMARDs and will be followed for an additional 15 months
- 6 months: discontinue vs continue DMARDs: (Protocol amendment 4.0)At 6 months, those patients still on Cimzia and DMARD therapy who were not randomized at month 3 AND achieve a change in DAS28> 1.2 will be randomized to discontinue versus continue DMARDs and will be followed for an additional 12 months.
- 6 months: D/C vs Cont'd DMARDs if change in DAS28: (Protocol amendment 4.0)At 6 months, if the change in DAS28 is at least 0.6 and there is a decision to continue Cimzia, then the patients will be randomized to discontinue versus continue DMARDs with Cimzia and will be followed for an additional 12 months.
- 3 or 6 months: stop CIMZIA and treat as per SOC: (Protocol amendment 4.0)If a change in DAS28 of <0.6 occurs at 6 months (at 3 months for protocol amendment 6.1)in patients not randomized at month 3 then the patient will stop Cimzia and treatment will be standard of care. However, patient will still be followed until the end of study.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of Cimzia given as an add-on to your current therapy with disease-modifying anti-rheumatic drug(s) (DMARDs)including MTX or given as monotherapy (alone) over an 18 month period.

Approximately 125 patients with moderate to severe Rheumatoid Arthritis (RA) who are being prescribed Cimzia will be enrolled into the study.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic systemic inflammatory disease that is associated with significant morbidity and mortality. The disease is characterized by inflammation of synovial joints that can result in pain, swelling and joint damage with secondary deformity and progressive disability and impairment of patient's health related quality of life. It is estimated that about 1% of the population worldwide has RA.

Treatment for RA includes use of nonsteroidal anti-inflammatory drugs (NSAIDs), cyclooxygenase-2 (COX-2) selective inhibitors, corticosteroids and DMARDs. The effectiveness and toxicities associated with use of DMARDs differs based on the individual agent; DMARDs are often partially effective. For those in whom DMARDs have not fully treated RA, TNF inhibitors are often prescribed.

TNFα plays an important role in RA. Activities ascribed to TNFα in RA include recruitment and activation of polymorphonuclear leukocytes (PMNs), cellular proliferation, increased prostaglandin and matrix-degrading protease activity, and bone and cartilage resorption.

CIMZIA (certolizumab pegol) in combination with methotrexate (MTX) is indicated for:

• reducing signs and symptoms, inducing major clinical response, and reducing the progression of joint damage as assessed by X-ray, in adult patients with moderately to severely active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 years of age.
2. Patient must be able to understand the information provided to them and to give written Informed Consent.
3. Patient must fulfill the old or new criteria for RA (see Appendix 1) or have a clinical diagnosis of RA.
4. Patient must be receiving (for 3 months before baseline) one of the following: methotrexate (≥ 12.5 mg) or another DMARD (leflunomide 10 to 20 mg/day, sulfasalazine >1000 mg/day, IM myochrysine for at least 20 weeks at 25 mg per month or more, azathioprine> 75mg/day), or combination DMARDs such as methotrexate with any other DMARD, or other combinations.
5. If patient is on prednisone they must be on a stable dose (≤ 10 mg/day) for 1 month prior to baseline.
6. Patient with active RA (≥ 3 SJC, on 28 joint count) who needs anti-TNF therapy as determined by the investigator and ability to obtain coverage for anti-TNF (Cimzia).
7. Patient must not have previously been exposed to Cimzia, however, previous anti-TNF exposure is allowed.
8. Patient with past anti-TNF exposure will be included if 1st anti-TNF was stopped due to secondary loss of efficacy, side effect or discontinuation for other reasons.
9. Patient must use Cimzia as per the dosing guidelines in the approved product monograph.

Exclusion Criteria:

1. Female patient who is breast-feeding or pregnant or does plan to become pregnant over the next year
2. Failure to use acceptable form of contraception in a pre-menopausal woman
3. Patient with concurrent serious liver disease
4. Patient with concurrent serious renal disease
5. Patient with significant hematological impairments
6. Patient with a history of cancer within the last 2 years, other than a successfully treated skin basal cell or squamous cell carcinoma and/or localized carcinoma in situ of the cervix
7. Patient with a history of malignant lymphoma of leukemia
8. Patient with a history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease (e.g. Multiple Sclerosis)
9. Patient with a history of untreated active tuberculosis
10. Patient with positive PPD (>5 mm) who have not had prophylaxis
11. Patient with a known positive HIV test
12. Patient with a persistent or severe infection(s) requiring hospitalization or treatment with iv antibiotics within 30 days or oral antibiotics within 7 days prior to baseline.
13. Patient with significant congestive heart failure
14. Patient with clinically significant concurrent medical of psychiatric disorders that in the physician's judgment may influence the study outcomes.
15. Patient with any condition that would prevent participation or completion in this study including language limitation or possibility that the patient will not be available for the complete study period
16. Patient with severe noncompliance
17. Patient receiving an experimental product within the last 6 weeks prior to first dose of Cimzia.
18. Other joint disease or joint pain condition where the patient or physician cannot distinguish RA assessments from the other joint disease
19. Concomitant SLE
20. Chest x-ray shows evidence of TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had not had an adequate response to a DMARD therapy will have Cimzia added to their existing DMARD therapy at baseline and will be followed.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-12; Primary Completion 2018-08-27 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients achieving DAS28<3.2 or maintaining a change in DAS from baseline of ≥ 1.2 at 18 months. | At 18 months
  Between-group differences with respect to the proportion of subjects achieving DAS28<3.2 will be assessed for statistical significance with the Chi-square test. Multiple-logistic regression model with terms for treatment group and potential confounders will be used to produce adjusted estimates of the relative rate of achieving therapeutic effectiveness. Time to achieving DAS28<3.2 will be assessed with Kaplan Meier survival analysis.

SECONDARY OUTCOMES:
Mean change from baseline in DAS28 score in each group at 18 months | At 18 months
  Between-group differences will be assessed for statistical significance with One Way ANOVA. General Linear Models will be used to adjust the between-group differences for potential confounders identified during the assessment of the baseline and demographic characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Pope, MD, Principal Investigator — Pope Research Corporation
Locations (13):
- Canada (13):
  - Rhumatologie Moncton, Moncton, New Brunswick
  - Eric N. Grant Professional Corp., Quispamsis, New Brunswick
  - Bowmanville, Ontario
  - Dr.'s Nalin and Vandana Ahluwalia Medicine Professional Corp., Brampton, Ontario
  - Brockville Medical Centre, Brockville, Ontario
  - The Arthritis Center, Burlington, Ontario
  - St. Joseph's Health Care, Guelph, Ontario
  - St-Joseph Health Center, London, Ontario
  - N.R. Medical Clinic, Markham, Ontario
  - Arthur Karasik Medicine Professional Corporation, Toronto, Ontario
  - Institut de Rhumatologie de Montréal, Montreal, Quebec
  - G.R.M.O. (Groupe de recherche en maladies oseuses) Inc., Québec, Quebec
  - Centre de Rhumatologie St-Louis, Québec, Quebec